CLINICAL TRIAL: NCT04109716
Title: School Adolescent Mood Project: Efficacy of IPT-AST in Schools
Acronym: SAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Institute of Education Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-016323; R305A190088 (Other Grant/Funding Number: U.S. Department of Education)
Record Dates: First submitted 2019-09-24; First posted 2019-09-30 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interpersonal Psychotherapy-Adolescent Skills Training (Experimental): Interpersonal Psychotherapy-Adolescent Skills Training (IPT-AST) is an indicated group depression prevention program. In IPT-AST, adolescents learn communication (e.g., using I statements, striking while the iron is cold) and interpersonal problem-solving strategies and apply these strategies to their relationships to decrease conflict, increase social support, and improve overall social functioning. IPT-AST consists of 1 or 2 individual pre-group sessions, 1 mid-group session, 8 weekly group sessions, and up to 6 individual booster sessions. Parents are invited to attend the mid-group session so the adolescents can apply the interpersonal strategies in a conversation with a parent. The purpose of the booster sessions is to monitor symptoms and apply the interpersonal strategies to current stressors. These sessions are designed to help solidify the interpersonal skills and address current problems before they result in a worsening of symptoms.
  Interventions: Behavioral: Interpersonal Psychotherapy - Adolescent Skills Training
- Services as Usual (SAU) (Active Comparator): Investigators anticipate that counselors in SAU will see youth in the study for brief, periodic sessions and/or will refer youth for treatment in the community. Counselors will be permitted to see the adolescents as often as they would like throughout the course of the study (up to 15-months post-baseline). Investigators will ask counselors to complete a form each time they see a teen, noting the length of the session, whether the session was scheduled or not, and the topics discussed.
  Interventions: Behavioral: Services as usual

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy - Adolescent Skills Training — This is an indicated group depression prevention consisting of 2 individual pre-group sessions, 8 weekly group session, and up to 6 individual booster sessions. IPT-AST will be delivered predominately through telehealth.
  Arms: Interpersonal Psychotherapy-Adolescent Skills Training
Behavioral: Services as usual — Services as usual is expected to be brief periodic sessions (in person or remote) with the school counselor or services in the community.
  Arms: Services as Usual (SAU)

SUMMARY:
This school-based randomized controlled trial will: a) examine the effects of telehealth-administered Interpersonal Psychotherapy-Adolescent Skills Training (IPT-AST), an evidence-based depression prevention program, as compared to services as usual (SAU) on social processes and emotional and school outcomes, b) examine moderators and mediators of intervention effects, and c) assess the costs, cost-effectiveness, acceptability, feasibility, fidelity, and sustainability of IPT-AST.

DETAILED DESCRIPTION:
This is a randomized clinical trial. Adolescents with elevated depressive symptoms will be identified and randomly assigned to IPT-AST delivered through telehealth by research staff (alone or in collaboration with school support staff) or services as usual (SAU) as delivered by counselors or other student support staff in schools. The research team will use longitudinal data collection with adolescents, parents, and counselors, and will collect data from teachers and school records to achieve study objectives.

Participants will be 240 racially and ethnically diverse students in the 9th and 10th grades between the ages of 14 and 17 with elevated symptoms of depression and their parents. Counselors in local high schools will also be study participants. A subset of counselors, adolescents, and administrators will also participate in a qualitative interview as part of an implementation study.

Adolescent participants will be randomly assigned to IPT-AST, an evidence-based depression prevention program, or SAU which may include supportive counseling and/or referral for services.

Standardized measures for adolescents, parents, and teachers and school records will be used to examine emotional outcomes (e.g., depression and anxiety symptoms, depression diagnoses) and school outcomes (e.g., school engagement, grades). Investigators will utilize standardized measures to assess social processes (e.g., interpersonal conflict, social functioning) that may mediate the effects of the intervention on these emotional and school outcomes. Investigators will also collect data on services received in IPT-AST and SAU, techniques utilized in both conditions, and feasibility, acceptability, fidelity, sustainability, and costs of IPT-AST using session logs, time diaries, standardized measures, leader- and consultant-rated fidelity checklists, and qualitative interviews.

ELIGIBILITY:
Adolescent Participants

Inclusion Criteria:

1. Adolescents in 9th or 10th grade between the ages of 14 and 17
2. Adolescent must be English-speaking; parents must be English or Spanish-speaking
3. Parental/guardian permission (informed consent) and child assent/consent
4. A score of 16 or higher on the CES-D AND at least 2 threshold or subthreshold symptoms on the K-SADS-PL
5. Have access to a cellular phone, computer, and/or tablet and have internet access to complete the remote intervention and evaluations

Exclusion Criteria:

1. Less than 2 threshold or subthreshold symptoms on the K-SADS-PL
2. Significant current active suicidal ideation reported on the K-SADS-PL at the eligibility evaluation or suicide attempt in the past year reported on the K-SADS-PL at the eligibility evaluation
3. Significant cognitive or language impairments requiring placement in Special Education as reported by the parent or as evident in the eligibility evaluation
4. Youth may be excluded on a case-by-case basis if the eligibility/baseline evaluation suggests that the group program would not be appropriate (for, instance, in the case of significant behavioral problems in the baseline evaluation).

For Parent Participants

Inclusion Criteria:

1. Parents of students in 9th or 10th grade between the ages of 14 and 17 at one of the participating schools
2. English or Spanish-speaking or limited English proficiency with use of interpreter
3. Consent to participate
4. Have access to a phone, computer, and/or tablet to complete remote evaluations

Exclusion Criteria:

None

For Parent-Designated Adult Family Member Participants (in cases where parent asks a different family member to complete parent assessments)

Inclusion Criteria:

1. 18 years of age or older
2. Knows the adolescent well enough to answer questions about him/her
3. English or Spanish-speaking or limited English proficiency with use of interpreter
4. Consent to participate
5. Have access to a phone, computer, and/or tablet to complete remote evaluations

Exclusion Criteria:

None

For Counselor Participants

Inclusion Criteria:

1. Counselor at one of the participating high schools
2. Consent to participate
3. Have access to a phone, computer, and/or tablet to complete remote evaluations

Exclusion Criteria:

None

For Teacher and Administrator Participants

Inclusion Criteria:

1. Teacher or administrator at one of the participating high schools
2. Consent to participate in the qualitative interview
3. Have access to a phone, computer, and/or tablet to complete remote evaluations

Exclusion Criteria:

None

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Depression symptoms | Screen, baseline, 2 month, 3 month, 9 month, 15 month
  Change in depression symptoms will be measured by the Center for Epidemiologic Studies-Depression Scale (CES-D) which assesses the frequency of 20 depressive symptoms over the past week; CES-D scores range from 0 to 60 (scores of 16 or higher are considered elevated); higher scores indicate more depression symptoms
Impairment | Baseline, 2 month, 3 month, 9 month, 15 month
  Change in impairment will be measured by the Columbia Impairment Scale (CIS), 13-item scale of overall functioning; scores range from 0-52; a score of 15 or higher is considered elevated impairment; higher scores represent greater impairment
Onset of depression diagnoses | Eligibility, 15 month
  The onset of diagnoses/change in depression diagnoses during the study period from eligibility to the 15 month assessment will be assessed by the Schedule for Affective Disorders and Schizophrenia for School-Age Children (K-SADS-PL)
Change in academic grades | Baseline, 15 month
  Impact of the intervention on school grades will be examined by accessing school records and looking at change in grades from baseline to the 15 month assessment.
Change in school attendance | Baseline, 15 month
  Impact of the intervention on school attendance will be examined by accessing school records and looking at change in attendance from baseline through 15 months.

SECONDARY OUTCOMES:
Internalizing and externalizing symptoms | Baseline, 2 month, 3 month, 9 month, 15 month
  Changes in internalizing and externalizing symptoms will be assessed by the Pediatric Symptom Checklist (PSC-17), which will be completed by teens, parents, and teachers; there is a total score (range of 0-34), internalizing subscale (0-24), externalizing subscale (0-20), and attention problems subscale (0-24); higher scores indicate more symptoms
Anxiety symptoms | Baseline, 2 month, 3 month, 9 month, 15 month
  Change in anxiety symptoms will be assessed by the Screen for Child Anxiety Related Disorders (SCARED), a 41-item scale assessing symptoms corresponding to different anxiety disorders; we will examine total scores and the following subscales: panic, GAD, and social anxiety; total scores range from 0-82 (25 or higher indicates clinical range); panic scores range from 0-26 (7 or higher indicates clinical range); generalized anxiety disorder scores range from 0-18 (scores of 9 or higher indicates clinical range); social anxiety scale ranges from 0-14 (scores 8 or higher indicate clinical range)
Number of disciplinary incidents | Baseline, 15 month
  Impact of the intervention on school disciplinary incidents will be examined by accessing school records and looking at number of new disciplinary incidents from baseline to the 15 month assessment
School connectedness | Baseline, 3 month, 9 month, 15 month
  Changes in school connectedness will be measured by the Psychological Sense of School Membership Scale, an 18 item measure of school connectedness; scores range from 18-90; higher scores indicate higher school connectedness
Emotional and behavioral engagement in learning | Baseline, 3 month, 9 month, 15 month
  The short and long-term impact of the interventions on engagement in learning will be measured by change in the Engagement versus Disaffection with Learning measure, a 20-item scale that assesses emotional and behavioral engagement vs. disengagement in school; total scores range from 20 to 80; behavioral and emotional engagement scores range from 10 to 40, with higher scores indicating greater engagement
Fidelity to the intervention | Weekly during intervention delivery
  The IPT-AST Fidelity Checklist will be completed by counselors and consultant to rate fidelity to IPT-AST intervention; adherence in each session is rated as a percent adherent; quality of session is also rated as percent; higher scores indicate greater adherence and quality (implementation)
Acceptability - counselors: A self-report measure, Counselor Feedback Form | 3 month, 15 month
  A self-report measure, Counselor Feedback Form, will be completed by any counselors who co-lead IPT-AST to assess acceptability of IPT-AST following group (3 month) and booster sessions (15 month) (implementation)
Acceptability - adolescents: A self-report measure, the Attitude Towards Intervention Questionnaire (ATI) | 3 month, 15 month
  A self-report measure, the Attitude Towards Intervention Questionnaire (ATI), will be completed by adolescents to assess acceptability of IPT-AST following group (3 month) and booster sessions (15 month) (implementation)
Patterns in qualitative data | 3 month
  Qualitative interviews will be conducted with IPT-AST stakeholders to gather information on implementation of IPT-AST; this is a qualitative interview which will be coded for key themes
Attendance | Weekly during IPT-AST
  Logs will track youth participation in IPT-AST and clinician attendance to IPT-AST consultation as one indicator of feasibility (implementation)

OTHER OUTCOMES:
Perspective-taking | Baseline, 2 month, 3 month, 9 month, 15 month
  Changes in perspective taking will be measured by the Interpersonal Reactivity Index (IRI), a 7-item perspective-taking scale; scores range from 0-28 with higher scores representing more perspective taking (social processes/mediators)
Social functioning | Baseline, 2 month, 3 month, 9 month, 15 month
  Changes in social functioning will be assessed by the Social Adjustment Scale-Self Report (SAS-SR), a 23-item scale of functioning in school (scores range from 6-30), with friends (scores range from 9-45), with family (scores range from 6-30), and dating (scores range from 2-10); a total score can also be computed (scores range from 23-115); higher scores indicate more difficulties in social functioning (social processes/mediators)
Quality of relationships: Inventory of Parent and Peer Attachment (IPPA-45) | Baseline, 2 month, 3 month, 9 month, 15 month
  Change in quality of relationships will be assessed by the Inventory of Parent and Peer Attachment (IPPA-45), a measure assessing the quality of mother (scores range from 15-75), father (scores range from 15-75), and peer relationships (scores range from 15-75); higher scores indicate more positive relationships (social processes/mediators)
Parent-child conflict | Baseline, 2 month, 3 month, 9 month, 15 month
  Changes in parent-child conflict will be assessed by the Conflict Behavior Questionnaire (CBQ), a 20-item questionnaire measuring conflict and negative communication between parents and adolescents; score range from 0-20; higher scores indicate more conflict (social processes/mediators)

CONTACTS AND LOCATIONS:
Overall Officials: Jami Young, PhD, Principal Investigator — CHOP, University of Pennsylvania Perelman School of Medicine
Locations (1):
- Children's Hopsital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The raw data will be entered into a de-identified electronic database and double-checked for accuracy. After data cleaning and quality assurance procedures are completed, pertinent sets of data will be converted into analytic datasets for statistical analyses. Additional variables may be derived for data analysis purposes. The cleaned, de-identified dataset, including additional derived variables, will be made accessible per IES data access requirements at the time that findings are published in a peer-reviewed journal. Data will be available for 10 years from that time.
Supporting Information: Study Protocol, ICF
Time Frame: The cleaned, de-identified dataset, including additional derived variables, will be made accessible per IES data access requirements at the time that findings are published in a peer-reviewed journal. Data will be available for 10 years from that time.
Access Criteria: Individuals interested in using the data should contact Dr. Young to make a request. Only de-identified data will be shared.

REFERENCES:
- [Derived] Young JF, Jones JD, Schwartz KTG, So A, Dysart GC, Kanine RM, Gillham JE, Gallop R, Davis M. Telehealth-delivered depression prevention: Short-term outcomes from a school-based randomized controlled trial. J Consult Clin Psychol. 2025 Apr;93(4):213-225. doi: 10.1037/ccp0000913. Epub 2024 Oct 31. PMID 39480285